CLINICAL TRIAL: NCT03565848
Title: Analysis of Surgical Outcomes in Women Undergoing Mesenteric Vascular and Nerve Sparing Surgery in Laparoscopic Segmental Colorectal Resection for Deep Infiltrating Endometriosis
Brief Title: Mesenteric Sparing Surgery in Laparoscopic Colorectal Resection for Endometriosis
Acronym: IRE-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Other Study IDs: IRE-1
Record Dates: First submitted 2018-05-30; First posted 2018-06-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Endometriosis; Bowel Endometriosis; Constipation
Keywords: Laparoscopy; Colorectal resection; Deep infiltrating endometriosis; Constipation
MeSH Terms: conditions — Endometriosis; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women underwent colorectal resection for endometriosis: Women referred for colorectal resection for deep infiltrating endometriosis that underwent laparoscopic segmental colorectal resection performed with mesenteric vascular and nerve sparing surgery.
  Interventions: Procedure: Mesenteric vascular and nerve sparing surgery in laparoscopic segmental colorectal resection

INTERVENTIONS:
Procedure: Mesenteric vascular and nerve sparing surgery in laparoscopic segmental colorectal resection — Laparoscopic segmental colorectal resection performed by dissecting adherent to the intestinal wall with mesenteric vascularization and innervation entirely preserved.

SUMMARY:
Colorectal resection is a standard surgical treatment of bowel deep infiltrating endometriosis (DIE). Nevertheless, concerns about different bowel functional outcomes related to radical surgery versus conservative surgery as shaving technique is a topic leading to much debate. Different surgical approach are used to perform colorectal resection and there is not a standardized technique. For the same concerns, studies have addressed the mesenteric vascular and nerve preservation both in oncological and benign intestinal disease with improved functional outcome. Therefore, the aim of this prospective study is to analyze feasibility and safety of mesenteric vascular and nerve Sparing Surgery in laparoscopic segmental colorectal resection for DIE with short and long term follow up. Women with DIE ,that underwent laparoscopic segmental colorectal resection, will undergo resection performed with inferior mesenteric artery and branching arteries preservation by dissecting adherent to the intestinal wall with mesenteric vascularization and innervation entirely preserved. Personal history, clinical data, surgical data, short and long term surgical complications and long term outcomes will be recorded. Symptoms and bowel function will be evaluated before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for bowel endometriosis requiring colorectal resection

Exclusion Criteria:

* None

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with deep infiltrating endometriosis underwent laparoscopic surgery treatment with segmental intestinal resection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in endometriosis related dysmenorrhea evaluated by Numeric Rating Scale for Pain | Change from baseline dysmenorrhea at 60 days after surgery and at 1 year after surgery
  Dysmenorrhea in 0 - 10 range according to the Numeric Rating Scale for Pain
Change in endometriosis related dyschezia evaluated by Numeric Rating Scale for Pain | Change from baseline dyschezia at 60 days after surgery and at 1 year after surgery
  Dyschezia in 0 - 10 range according to the Numeric Rating Scale for Pain
Change in endometriosis related dyspareunia evaluated by Numeric Rating Scale for Pain | Change from baseline dyspareunia at 60 days after surgery and at 1 year after surgery
  Dyspareunia in 0 - 10 range according to the Numeric Rating Scale for Pain.
Change in endometriosis related dysuria evaluated by Numeric Rating Scale for Pain | Change from baseline dysuria at 60 days after surgery and at 1 year after surgery
  Dysuria in 0 - 10 range according to the Numeric Rating Scale for Pain.
Change in endometriosis related pelvic chronic pain evaluated by Numeric Rating Scale for Pain | Change from baseline pelvic chronic pain at 60 days after surgery and at 1 year after surgery
  Pelvic chronic pain in 0 - 10 range according to the Numeric Rating Scale for Pain.
Change in bowel symptoms evaluated by Constipation Assessment Scale | Change from baseline bowel symptoms at 60 days after surgery and at 2 year after surgery
  Bowel symptoms in 0 - 16 range according to the Constipation Assessment Scale. Constipation Assessment Scale includes eight items, each of which is self-rated by the patient as 'no problem' (score of 0), 'some problem' (score of 1), or 'severe problem' (score of 2). The item ratings are then summed, so the overall score may range from 0 (no constipation) to 16 (worst possible constipation).

SECONDARY OUTCOMES:
Endometriosis characteristics | intraoperative
  rAFS classification
Complication rate | Within 6 months after surgery
  Number of surgical complications (Clavien-Dindo Classification)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Garzon, M.D., Principal Investigator — Universita di Verona; Antonio Simone Laganà, M.D., Principal Investigator — Uninsubria; Paola Pomini, M.D., Principal Investigator — Universita di Verona; Massimo Franchi, M.D., Principal Investigator — Universita di Verona

IPD SHARING:
Plan to Share IPD: Undecided